CLINICAL TRIAL: NCT00414336
Title: Randomized, Controlled, Phase 1 Study of the Safety and Immunogenicity of the AMA1-C1/Alhydrogel + CPG 7909 Vaccine for Plasmodium Falciparum Malaria in Semi-Immune Malian Adults
Brief Title: Phase I Study of Safety and Immunogenicity of AMA1-C1Alhydrogel + CPG 7909 Vaccine for Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases@@@Coley Pharmaceutical Group (Unknown)
Responsible Party: RCHSPB
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 999907051; 07-I-N051
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-04

CONDITIONS: Malaria
Keywords: Blood Stage; Investigational; Endemic; Malaria
MeSH Terms: conditions — Malaria; Burkitt Lymphoma

INTERVENTIONS:
Drug: AMA1-C1/Alhydrogel + CPG 7909 Vaccine

SUMMARY:
This study will evaluate the safety of an experimental vaccine can protect people from malaria and study its effects. Malaria, which affects many people in Mali and other countries in Africa, is caused by germs spread by mosquito bites. In Mali, the disease is the leading cause of death. Researchers at the Malaria Research and Training Center at the University of Bamako are working with NIH to develop an experimental vaccine against the disease. The vaccine, called AMA1-C1Alhydrogel (or AMA1-C1), contains a small part of the malaria-causing germ. CPG-7909 is a product to improve the body's reactions to vaccines.

Patients ages 18 to 45 who are in good health, who live in Don gu bougou, Mali, and plan to stay there for the study duration, and who are not pregnant or breast feeding may be eligible for this study. There will be 24 participants.

At an initial evaluation of 2 to 3 hours, patients will have a physical examination and undergo blood and urine tests regarding the blood, kidneys, and liver. During the study, patients will receive two injections of one of the two experimental malaria vaccines. Injections of the same vaccine each time, 4 weeks apart, are given in an arm muscle. Patients will receive either AMA1-C1 or AMA1-C1 with CPG-7909 but will not know which of the vaccines they receive until the study's end. After each injection, patients will stay in the clinic for 30 minutes for observation. They will return after 1, 2, 3, 7, and 14 days to be examined and report how they are feeling. Blood and urine samples will be collected at some visits. Each clinic visit takes 1 to 2 hours. If for some reason a patient receives only one injection, he or she will be asked to return to the clinic for routine visits until the study's end. After the first 2 months, patients will return to the clinic once a month for 30 weeks. In that period, 12 blood samples will be taken. Researchers want to be sure that the vaccine is not harmful as well as to measure the vaccine's effects.

Risks in this study include pain, swelling, and redness at the injection site; fever; and gastrointestinal problems. Some people have had a temporary decrease in white blood cells after receiving the vaccine. There is a small chance of a severe allergic reaction. However, researchers will closely watch patients immediately after each injection and will give treatment if a serious reaction occurs.

Participants will receive 75 kilos of rice and 75 kilos of millet (165 lb. of ...

DETAILED DESCRIPTION:
AMA1-C1 + CPG 7909 is a blood stage malaria vaccine candidate. The primary objective of this Phase 1 study is to evaluate safety and reactogenicity of the vaccine in semi-immune adults in Mali. Secondary objectives are to evaluate the immunogenicity of the vaccine. The study is a double blind Phase 1 clinical trial in healthy adult volunteers. Volunteers will be screened and 24 participants will be enrolled and randomly assigned to one of the two groups: 12 volunteers will receive two doses of 80 microgram AMA1-C1/Alhydrogel + 500 microgram CPG; 12 volunteers will receive 80 microgram AMA1-C1/Alhydrogel, both at a 1-month dosing interval. Safety outcome measures are local and systemic (including laboratory) adverse events. Immune responses to vaccination will be measured by enzyme-linked immunosorbent assay (ELISA) and growth inhibition assay (GIA), and will be compared between groups. Peripheral blood lymphocytes will be assayed for the presence of AMA-1-specific memory B cells and for the total number of memory B cells.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males or females between 18 and 45 years, inclusive.
  2. Known residents of the village of Don gu bougou, Mali.
  3. Good general health as determined by means of the screening procedure.
  4. Available for the duration of the trial (30 weeks).
  5. Willingness to participate in the study as evidenced by signing the informed consent document.

EXCLUSION CRITERIA:

1. Pregnancy as determined by a positive urine beta-hCG at any point during the study (if female).
2. If female, participant and her spouse have not used or are unwilling to use reliable contraceptive methods such as: abstinence, birth control pills or birth control patches or vaginal ring, diaphragm with spermicide, IUD (intrauterine device), condom with spermicide, progestin implant or injection, or surgical sterilization (hysterectomy, bilateral oophorectomy, tubal ligation) prior to enrollment to 3 months after the second vaccination. (At the time of vaccination a female participant must have a negative urine pregnancy test on two occasions at least two weeks apart, and must have used a reliable contraceptive method in the interim).
3. Currently lactating and breast-feeding (if female).
4. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, chronic infectious or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
5. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.
6. Pre-existing known autoimmune diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia.
7. Laboratory evidence of possible autoimmune disease determined by anti-dsDNA titer that equals or exceeds 25 IU.
8. Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25 times the upper limit of normal of the testing laboratory).
9. Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory, or more than trace protein or blood on urine dipstick testing confirmed by repeat testing of clean-catch, midstream sample). (More than trace blood on urine dipstick will not exclude a female who is actively menstruating.)
10. Laboratory evidence of hematologic disease (absolute leukocyte count less than 3000/mm(3) or greater than 11,500/mm(3); hemoglobin less than 0.9 times the lower limit of normal of the testing laboratory, by gender; absolute granulocyte count less than 1300/ mm(3); absolute lymphocyte count less than 1000/mm(3); or platelet count less than 110,000/mm(3)).
11. Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
12. Participation in another investigational vaccine or drug trial within 30 days of starting this study, or while this study is ongoing.
13. Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
14. History of a severe allergic reaction or anaphylaxis.
15. Severe asthma. This will be defined as:

    * Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or parenteral corticosteroids;
    * Clinically significant reactive airway disease that does not respond to bronchodilators.
16. Positive rapid diagnostic test for anti-Hepatitis C virus (HCV).
17. Positive rapid diagnostic test for Hepatitis B surface antigen (HBsAg).
18. Known immunodeficiency syndrome.
19. Use of systemic corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study.
20. Receipt of a live vaccine within past 4 weeks or a non-live vaccine within past 2 weeks prior to entry into the study.
21. History of a surgical splenectomy.
22. Receipt of blood products within the past 6 months.
23. Previous receipt of an investigational malaria vaccine.
24. History of a known allergy to nickel.
25. History of known allergy to yeast.
26. History of use of chloroquine or related compounds (amodiaquine or primaquine) within 8 weeks of study entry.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150
Dates: Start 2006-12-15; Primary Completion 2006-12-15 (Actual); Study Completion 2006-12-15 (Actual)

PRIMARY OUTCOMES:
Safety and reactogenicity.

SECONDARY OUTCOMES:
To determine the level and kinetics of the antibody response elicited by AMA1-C1/Alhydrogel + CPG

CONTACTS AND LOCATIONS:
Locations (1):
- Doneguebougou Malaria Vaccine Center, Donéguébougou, Mali

REFERENCES:
- [Background] Hodder AN, Crewther PE, Anders RF. Specificity of the protective antibody response to apical membrane antigen 1. Infect Immun. 2001 May;69(5):3286-94. doi: 10.1128/IAI.69.5.3286-3294.2001. PMID 11292751
- [Background] Malkin EM, Diemert DJ, McArthur JH, Perreault JR, Miles AP, Giersing BK, Mullen GE, Orcutt A, Muratova O, Awkal M, Zhou H, Wang J, Stowers A, Long CA, Mahanty S, Miller LH, Saul A, Durbin AP. Phase 1 clinical trial of apical membrane antigen 1: an asexual blood-stage vaccine for Plasmodium falciparum malaria. Infect Immun. 2005 Jun;73(6):3677-85. doi: 10.1128/IAI.73.6.3677-3685.2005. PMID 15908397
- [Background] Cooper CL, Davis HL, Morris ML, Efler SM, Adhami MA, Krieg AM, Cameron DW, Heathcote J. CPG 7909, an immunostimulatory TLR9 agonist oligodeoxynucleotide, as adjuvant to Engerix-B HBV vaccine in healthy adults: a double-blind phase I/II study. J Clin Immunol. 2004 Nov;24(6):693-701. doi: 10.1007/s10875-004-6244-3. PMID 15622454